CLINICAL TRIAL: NCT07161778
Title: A Phase II Single Arm, Multi-centre Trial of Triamcinolone With a GnRH Analog for Castration Resistant Prostate Cancer
Brief Title: A Trial of Triamcinolone With a GnRH Analog for Castration Resistant Prostate Cancer
Acronym: TRICREST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7664; 2010-022010-32 (EudraCT Number)
Record Dates: First submitted 2014-10-21; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Castration Resistant Prostate Cancer
Keywords: CRPC
MeSH Terms: interventions — Triamcinolone Acetonide; Injections, Intramuscular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triamcinolone (Experimental): An initial loading dosage will be given and then every 4 weeks the patient will be given triamcinolone. Triamcinolone acetonide IM injection should be administered as per individual sites local procedures.
  The number of Triamcinolone injections, the volume and the site of administration will be documented in the CRF. The initial dose can be split according to local administration procedures.
  Cycle 1
  Day 1 Week 1 (loading dose given once only)
  o 360 mg IM injection
  Subsequent cycles (given 4 weekly thereafter until progression +/-3 days)
  Day 1
  o 120 mg IM injection
  Interventions: Drug: Triamcinolone acetonide IM injection

INTERVENTIONS:
Drug: Triamcinolone acetonide IM injection — An initial loading dosage will be given and then every 4 weeks the patient will be given triamcinolone. Triamcinolone acetonide IM injection should be administered as per individual sites local procedures.
  The number of Triamcinolone injections, the volume and the site of administration will be documented in the CRF. The initial dose can be split according to local administration procedures.
  Cycle 1
  Day 1 Week 1 (loading dose given once only)
  o 360 mg IM injection
  Subsequent cycles (given 4 weekly thereafter until progression +/-3 days)
  Day 1
  o 120 mg IM injection
  Other Names: Kenalog Intra-articular / Intramuscular Injection

SUMMARY:
When metastatic prostate cancer becomes unresponsive to hormone therapy, it is known as castration resistant prostate cancer, treatment options are limited and response to this treatment can be short.

The standard treatment for this type of cancer (hydrocortisone or dexamethasone) gives an average response time of 4 months. After this chemotherapy would be considered. In this patient population the majority of men are aged over 70, so giving chemotherapy with its associated toxicities; can reduce the quality of life for patients, and it is preferable to delay this treatment option until absolutely necessary. With this in mind, treating with triamcinolone aims to increase this period of response.

One of the ways that castration resistant prostate cancer develops is by acquiring a mutations that allow it to respond to other steroids both endogenous e.g. cortisol and also to synthetic steroids being used to control the disease e.g. dexamethasone. No known mutation allows a response to triamcinolone, a unique finding amongst steroids.

To date there has been one clinical study looking at giving oral triamcinolone, but as yet there has been not study of intramuscular triamcinolone

DETAILED DESCRIPTION:
Castration resistant prostate cancer (CRPC) is a cancer which has become resistant to hormone therapy. Triamcinolone is a steroid drug, and it is hoped that when administered intra-muscularly with a gonadotropin-releasing hormone (GnRH) analog, it will reduce the tumours' ability to grow and thus improve the therapy response rate.

This is a single arm, multi-centre phase II trial and it follows a Simon Two-stage minimax design based on the progression free survival rate at 6-months. A total of 41 patients will be recruited to the study. Following recruitment of the first 17 patients; an interim analysis will take place, and at least 7 of these will be required to have survived progression free, at 6 months in order to proceed to the 2nd stage of the trial. During the 2nd stage, if 20 or more patients out of the total 41 have survived progression free, then the drug will be developed further at a randomized phase II or phase III trial.

Patients will receive monthly treatment of intramuscular triamcinolone and GnRH up until treatment failure (progression, toxicity or death) and survival information will then be collected.

Patients will be identified through referrals and at multidisciplinary team meetings (MDTs). Eligible patients will be approached by members of the research team at outpatient clinic appointments. To be registered, the trial patients must satisfy all aspects of the eligibility criteria.

Once an eligible patient is identified and prior to their participation in this study, the Investigator, or a person delegated by the Investigator will adequately explain the aims, methods, anticipated benefits, potential hazards, and relay the fact that should new safety information result in significant changes in the risk or benefit, study patients will be notified. The Investigator, or a person delegated by the Investigator must also explain to the patient that they are completely free to refuse to enter the study or to withdraw at any time during the study. The patient will be sent away with a patient information sheet and will be given at least 24 hours to consider study participation.

If the eligible patient is satisfied and fully understands what the study entails and what is expected, written informed consent will be obtained and the patient will be registered into the trial. A blood test will be taken at 9am in the morning; the equivalent of 3 teaspoons of blood will be removed. The blood test will be used to assess blood circulating tumour cells (CTC), toxicity tumour markers, and the levels of cortisol and protein specific antigen (PSA is a chemical prostate cancer produces). A full history will be taken, and the patient will be examined. A bone scan performed prior to study participation as part of standard practice will also be assessed, providing it is not dated beyond a maximum of 6 weeks prior to the start of trial treatment. The inclusion and exclusion criteria will be verified once more.

One day one, week one of treatment, the patient will be asked to return a 24 hour urine collection sample ( in order to obtain a profile of urinary steroids). The patient will receive an initial loading dose of 360 mg of triamcinolone, this will be administered over 3 injections (3 x 120 mg) into the muscle in the patient's buttocks. On day one, week four of treatment, the patient will receive only one injection of 120 mg IM of triamcinolone, and thereafter there will be one injection per treatment visit, four weekly until progression (as per day one, week four of treatment).

Depending on the GnRH analog treatment the patient was on prior to the start of the trial, either 4 weekly or 12 weekly, it will remain the same for the duration of the patient's participation in the trial. The GnRH analog can be administered by their local GP as custom or if they are due receive the GnRH analog and triamcinolone at the same time, both will be administered at the site. However triamcinolone can be administered at the site only.

The patient will be monitored with a follow up phone call from a nurse within a week following the first loading dose of triamcinolone, to see how the patient is and to check if there are any side-effects of the treatment.

Three weeks following the start of treatment a blood test and 24-hour urine collection will be repeated. This is to assess whether the cancer is responding to treatment. These tests are also scheduled to be performed when the patient attends 4 weekly for triamcinolone treatment, however the doctor may request further tests depending on how the patient is responding to treatment. In particular, if PSA increases significantly while on treatment, the doctor may then decide to stop triamcinolone treatment and inform the patient of alternative treatment options. Following treatment failure, patients will be followed up every 3 months and permission will be sought to obtain patient survival data when they return to standard care appointments.

An additional aspect of the study which is optional depending on the site and the patient is the translational research component:

Provided the patient has not withheld consent, a blood sample will be taken at the start of the trial, following registration and another sample when treatment fails due to progression, which will then be used to analyse DNA mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate
2. Progressive disease despite castration with an elevated PSA >5ng/ml (testosterone <1.5nmol/l or failure of GnRH analogue with peripheral anti-androgen if non-castrate level on GnRH alone)
3. ECOG performance status (PS) 0-3 and considered by responsible consultant suitable to undergo treatment
4. Males aged greater or equal than 18
5. Patients who are able to understand their participation in the study and give written informed consent

Exclusion Criteria:

1. Contraindication to intramuscular injections
2. Unable to titrate medication for type 2 diabetes if deterioration in control on triamcinolone
3. Absolute contraindication to corticosteroids
4. Previous use of corticosteroids in prostate cancer
5. Previous chemotherapy for prostate cancer
6. Current participation in any other investigational drug study
7. History of a malignancy within 5 years except those treated with curative intent for skin cancer (other than melanoma)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-10-19 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Progression free survival in patients with CRPC | 6 months
  To examine whether triamcinolone (IM injection) offers an increased progression free survival (PFS) in patients with confirmed CRPC.

SECONDARY OUTCOMES:
Time to PSA progression according to PCWG2 | Measured at the beginning of every treatment cycle (Time to PSA progression from baseline - 6 month)
  Serum collected will be tested for PSA progression
Circulating Tumour Cells response in patients after 28 days of treatment | Circulating Tumour Cells results at baseline and taken 28 days post baseline will be compared
  Comparing CTC at baseline to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shamash, MD FRCP, Principal Investigator — Barts & The London NHS Trust
Locations (3):
- United Kingdom (3):
  - Royal Sussex County Hospital, Brighton
  - Raigmore Hospital, Inverness
  - St Bartholomew's Hospital, London

REFERENCES:
- [Background] Buchanan G, Yang M, Harris JM, Nahm HS, Han G, Moore N, Bentel JM, Matusik RJ, Horsfall DJ, Marshall VR, Greenberg NM, Tilley WD. Mutations at the boundary of the hinge and ligand binding domain of the androgen receptor confer increased transactivation function. Mol Endocrinol. 2001 Jan;15(1):46-56. doi: 10.1210/mend.15.1.0581. PMID 11145738
- [Background] Marcelli M, Ittmann M, Mariani S, Sutherland R, Nigam R, Murthy L, Zhao Y, DiConcini D, Puxeddu E, Esen A, Eastham J, Weigel NL, Lamb DJ. Androgen receptor mutations in prostate cancer. Cancer Res. 2000 Feb 15;60(4):944-9. PMID 10706109
- [Background] Chang CY, Walther PJ, McDonnell DP. Glucocorticoids manifest androgenic activity in a cell line derived from a metastatic prostate cancer. Cancer Res. 2001 Dec 15;61(24):8712-7. PMID 11751389
- [Background] Zhao XY, Malloy PJ, Krishnan AV, Swami S, Navone NM, Peehl DM, Feldman D. Glucocorticoids can promote androgen-independent growth of prostate cancer cells through a mutated androgen receptor. Nat Med. 2000 Jun;6(6):703-6. doi: 10.1038/76287. PMID 10835690
- [Background] Srinivas S, Krishnan AV, Colocci N, Feldman D. Phase II study evaluating oral triamcinolone in patients with androgen-independent prostate cancer. Urology. 2006 May;67(5):1001-6. doi: 10.1016/j.urology.2005.11.004. PMID 16698360
- [Background] Ogirala RG, Aldrich TK, Prezant DJ, Sinnett MJ, Enden JB, Williams MH Jr. High-dose intramuscular triamcinolone in severe, chronic, life-threatening asthma. N Engl J Med. 1991 Feb 28;324(9):585-9. doi: 10.1056/NEJM199102283240903. PMID 2021388
- [Background] McGivney SA, Ogirala RG. Effect of high-dose intramuscular triamcinolone in older adults with severe, chronic asthma. Lung. 1994;172(2):73-8. doi: 10.1007/BF00185078. PMID 8114514
- [Background] Veldscholte J, Berrevoets CA, Ris-Stalpers C, Kuiper GG, Jenster G, Trapman J, Brinkmann AO, Mulder E. The androgen receptor in LNCaP cells contains a mutation in the ligand binding domain which affects steroid binding characteristics and response to antiandrogens. J Steroid Biochem Mol Biol. 1992 Mar;41(3-8):665-9. doi: 10.1016/0960-0760(92)90401-4. PMID 1562539
- [Background] Ross RW, Oh WK, Xie W, Pomerantz M, Nakabayashi M, Sartor O, Taplin ME, Regan MM, Kantoff PW, Freedman M. Inherited variation in the androgen pathway is associated with the efficacy of androgen-deprivation therapy in men with prostate cancer. J Clin Oncol. 2008 Feb 20;26(6):842-7. doi: 10.1200/JCO.2007.13.6804. PMID 18281655
- [Background] Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, Eisenberger MA, Higano C, Bubley GJ, Dreicer R, Petrylak D, Kantoff P, Basch E, Kelly WK, Figg WD, Small EJ, Beer TM, Wilding G, Martin A, Hussain M; Prostate Cancer Clinical Trials Working Group. Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008 Mar 1;26(7):1148-59. doi: 10.1200/JCO.2007.12.4487. PMID 18309951
- [Background] Shamash J, Powles T, Sarker SJ, Protheroe A, Mithal N, Mills R, Beard R, Wilson P, Tranter N, O'Brien N, McFaul S, Oliver T. A multi-centre randomised phase III trial of Dexamethasone vs Dexamethasone and diethylstilbestrol in castration-resistant prostate cancer: immediate vs deferred Diethylstilbestrol. Br J Cancer. 2011 Feb 15;104(4):620-8. doi: 10.1038/bjc.2011.7. Epub 2011 Feb 1. PMID 21285990
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- See also: Related Info — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2010-022010-32